CLINICAL TRIAL: NCT05081102
Title: A Clinical, Multicenter, Randomized, Parallel-group, Double-dummy, Comparative Study of Non-inferiority of the Fixed-dose Combination of Oxycodone 5 Mg/ibuprofen 400 Mg from Eurofarma Versus Tylex® (codeine 30 Mg/paracetamol 500 Mg) in the Treatment of Moderate to Intense Pain Post-impacted Third Lower Molar Extraction
Brief Title: Fixed-dose Combination of Oxycodone [OXIcodona] + IbuproFEN in Pain Relief After Third Molar Extraction
Acronym: OXIFEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF-176
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pain
Keywords: postoperative; third lower molar extraction
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: FDC oxycodone 5 mg/ibuprofen 400 mg from Eurofarma Laboratórios SA (experimental drug) (Experimental): Participants randomized to this group will receive one (01) tablet of the experimental drug + one (01) tablet of Tylex® placebo when post-surgical pain intensity reaches moderate to intense intensity (≥ 40 mm on a 0-100 mm VAS). Participants will be instructed to, from then on, use this same treatment whenever needed for pain relief, observing a minimum interval of six (06) hours between two intakes, for up to 3 days (72 hours after the initial dose).
  Interventions: Drug: FDC of oxycodone 5 mg/ibuprofen 400 mg
- Group 2: Tylex® (codeine 30 mg/paracetamol 500 mg) (Active Comparator): Participants randomized to this group will receive one (01) Tylex® tablet (codeine 30 mg/paracetamol 500 mg) + one (01) tablet of FCD placebo when post-surgical pain intensity reaches moderate to intense intensity (≥ 40 mm on a 0-100 mm VAS). Participants will be instructed to, from then on, use this same treatment whenever needed for pain relief, observing a minimum interval of six (06) hours between two intakes, for up to 3 days (72 hours after the initial dose).
  Interventions: Drug: Tylex

INTERVENTIONS:
Drug: FDC of oxycodone 5 mg/ibuprofen 400 mg — receive one (1) experimental drug tablet (FCD of oxycodone 5mg/ibuprofen 400mg) + one (1) Tylex® placebo.
  Arms: Group 1: FDC oxycodone 5 mg/ibuprofen 400 mg from Eurofarma Laboratórios SA (experimental drug)
Drug: Tylex — receive one (1) Tylex® tablet (codeine 30 mg/paracetamol 500 mg) + one (1) FDC placebo tablet
  Arms: Group 2: Tylex® (codeine 30 mg/paracetamol 500 mg)

SUMMARY:
A clinical, multicenter, randomized, parallel-group, double-blind, double-dummy, comparative study of non-inferiority.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil) .

DETAILED DESCRIPTION:
Patients aged between 16 and 35 years with indication for surgical removal of impacted lower third molar will be randomized at a 1:1 ratio to receive FDC oxycodone 5 mg/ibuprofen 400 mg from Eurofarma Laboratórios SA (experimental drug) or FDC codeine 30 mg/paracetamol 500 mg (Tylex® - Janssen-Cilag Farmacêutica Ltda.) as tablets, for up to three (03) days. Participants whose surgery lasts no more than 40 minutes (starting from the initial incision to the extraction of impacted third molar) and who experience post-surgical pain that is moderate to intense in intensity up to four (04) hours after the surgery ends will be randomized. The first administration of the study treatment will be performed at the clinical investigation site when post-surgical pain reaches moderate/intense intensity (≥ 40 mm on a 0-100 mm Visual Analogue Scale [VAS]).

Participants will be instructed to, from then on, use the study treatment as needed for pain relief, observing a minimum interval of six (06) hours between two intakes, for up to three (03) days (72 hours after the initial dose).

Subjects who meet all of the eligibility criteria will be randomized to one of the following treatment groups:

Group 1: FDC oxycodone 5 mg/ibuprofen 400 mg from Eurofarma Laboratórios SA (experimental drug) - Participants randomized to this group will receive one (01) tablet of the experimental drug + one (01) tablet of Tylex® placebo when post-surgical pain intensity reaches moderate to intense intensity (≥ 40 mm on a 0-100 mm VAS).

Group 2: Tylex® (codeine 30 mg/paracetamol 500 mg) - Participants randomized to this group will receive one (01) Tylex® tablet (codeine 30 mg/paracetamol 500 mg) + one (01) tablet of FCD placebo when post-surgical pain intensity reaches moderate to intense intensity (≥ 40 mm on a 0-100 mm VAS).

The subjects will be allowed to use the rescue medication if necessary:

Paracetamol 500 mg (Tylenol® 500 mg).

All subjects must have three (3) on-site visits at the research site. Three (3) phone calls will take place between the on-site visits: Screening visit (Vs), randomization visit (Vr), first phone call (CT1), second phone call (CT2), third phone call (CT3), final visit (Vf).

The period for enrolling participants in the study will begin after the necessary ethical and regulatory approvals and will have an estimated duration of up to 12 months.

The approximate duration of the study will be 16 ± 2 days for each participant.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 16 and 35 years old (inclusive).
2. Presence of impacted third lower molar with surgical removal indicated (diagnosed via panoramic x-ray within six [6] months before inclusion in the study), at vertical, mesioangular or horizontal position as per the Winter's classification, provided that it belongs to the following Pell & Gregory's classes.
3. Maximum surgery duration of 40 minutes, counted from the initial incision to the impacted third molar extraction.
4. Moderate to intense postoperative pain (≥ 40 mm at a VAS of 0-100 mm) up to four (4) hours after the end of the surgery (counted from the end of the suture).
5. Informed Consent Form (ICF) and Informed Assent Form (IAF) signature, when applicable, before performing any study procedure

Exclusion Criteria:

1. Known hypersensitivity to oxycodone or other opioid agents.
2. Known hypersensitivity to ibuprofen, acetylsalicylic acid (ASA), or any other non-steroidal anti-inflammatory drug (NSAID).
3. Known hypersensitivity to paracetamol or to any component of the Tylex® formulation;
4. History of bronchospasm or other anaphylactoid reactions (e.g.: hives, rhinitis, angioedema) associated with the use of analgesics, such as salicylates, paracetamol, diclofenac, ibuprofen, indomethacin, naproxen;
5. Abuse of illegal drugs, including alcoholism; emotional instability and/or previous attempt of suicide;
6. Pregnancy or breastfeeding.
7. Women of childbearing potential who do not agree to use a known effective birth control method, unless the participants are surgically sterile or state they are expressly free of the risk of getting pregnant for not having sexual intercourse or for having sexual intercourse with no reproductive potential.
8. Known hepatic or renal failure.
9. Participation in a clinical research protocol within the past 12 months, unless the investigator considers that the participation in the study could result in a direct benefit to the subject.
10. Presence of any condition that, in the investigator's opinion, would make the subject ineligible to participate in the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 288 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
sum of pain relief scores over 6 hours (TOTPAR6) | 6 hours
  After the administration of the first dose of study treatment, participants will assess pain relief using the 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) in one-hour intervals (1, 2, 3, 4, 5, and 6 h). The sum of pain relief scores within 6 hours determines TOTPAR6, which ranges from 0 to 24, and the higher the value, the greater the pain relief.

SECONDARY OUTCOMES:
Sum of pain relief scores over four (4) hours (TOTPAR4) | 4 hours
  After the first study treatment dose is given, subjects will evaluate the pain relief using a 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) in 1-hour intervals (1, 2, 3, 4 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No